CLINICAL TRIAL: NCT05782010
Title: SCI-Pex, a Multi-center, Prospective, Non-controlled Investigation to Evaluate the Safety and Performance of PexyEazy®, a Device for Treatment of Hemorrhoids
Brief Title: SCI-Pex Study - Safety and Performance of PexyEazy®, a Device for Treatment of Hemorrhoids
Acronym: SCI-Pex
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Developeration AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIV-23-01-041830
Record Dates: First submitted 2023-01-16; First posted 2023-03-23 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Hemorrhoids; Hemorrhoids, Internal; Suture; Complications, Infection or Inflammation; Rectal Diseases; Gastrointestinal Diseases
Keywords: PexyEazy
MeSH Terms: conditions — Hemorrhoids; Infections; Inflammation; Rectal Diseases; Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PexyEazy procedure (Experimental): PexyEazy procedure on patients with hemorrhoidal disease grade II and III. The study is descriptive and non-comparable to evaluate the safety and performance of PexyEazy.
  Interventions: Device: PexyEazy

INTERVENTIONS:
Device: PexyEazy — PexyEazy procedure on patients with hemorrhoidal disease grade II and III. The study is descriptive and non-comparable to evaluate the safety and performance of PexyEazy.

SUMMARY:
The SCI-Pex study is a multicenter, prospective, non-controlled investigation on PexyEazy®, a new device for treatment of hemorrhoids based on the mucopexy method. Mucopexy is a well established method where sutures are applied above the hemorrhoids. When knots are tied, the hemorrhoids are lifted inwards to their normal position, which makes them swell down and symptoms disappears. PexyEazy® perform a mukopexy in a semiautomatic, faster and easier way on awake patient in less than 10 minutes. The SCI-Pex study will evaluate the safety and performance of PexyEazy on 35 patients with hemorrhoids grade II and III with a follow-up after 1 week, 3 months and 1 years. Adverse events, pain and other complications will be recorded, quality of life and hemorrhoid symptom questionnaires and clinical examination after 3 months and 1 year will be monitored to evaluate the result after a PexyEazy® procedure.

DETAILED DESCRIPTION:
Background:

The generally accepted theory of why hemorrhoidal disease (HD) occurs is that the hemorrhoidal cushions slid down in the anal canal (muco-anal prolapse), which allows them to swell up. This creates problems with bleeding, leakage (soiling), itching and pain.

Traditionally, severe HD is treated by surgical removal of the hemorrhoids, but the procedure is associated with long recovery time, pain and complications like stenosis and incontinence. Minimal invasive and hemorrhoid preserving surgery has gained popularity during the last two decades with new methods like Procedure for Prolapse and Hemorrhoids (PPH)/Stapled Anopexy and Transanal Hemorrhoidal Dearterialisation (THD)/Hemorrhoidal Artery Ligation and Recto Anal Repair (HAL/RAR). Several studies have shown, thought that mucopexy alone result in equally good result as THD/HAL-RAR. There are several ways to perform a mucopexy with different ways in how the sutures are applied and how many rows of sutures that are done.

Other available methods focus on tissue destruction, for example sclerosing injections, laser, radio ablation, or methods with applied electricity that induce heat. These methods make the hemorrhoids to swell down but does not treat the muco-anal prolapse that are present in grade II and III hemorrhoids.

PexyEazy® perform a mucopexy in a new, semi-automatic way with the benefit of reducing the cost and time of surgery and is estimated to be able to be conducted without the need of general anesthesia.

Method:

PexyEazy® is a single-use device for surgical treatment of internal HD grade II and III (according to the Goligher classification). It is based on the mucopexy method, but instead of applying the sutures by hand, the mucosa is folded by the device and then a loop of suture is introduced into the folded mucosa. When knots are applied, the hemorrhoids are lifted inwards, as the folded mucosa above the hemorrhoids is pulled together. Due to that the most proximal suture is longer and deeper and acts as an anchoring stich, the lifting motion is inwards, towards the deeper stitch. When the position of the hemorrhoids is normalized, the venous drainage is improved, and the hemorrhoids swell down, and symptoms disappears.

PexyEazy® consists of five major parts: PexyEazy® examination proctoscope, handle with depth setting piston, light shuttle with a led lamp, PexyEazy® Mucopexy Device (MD) and the battery-pack. All parts are sterile, except the re-usable battery-pack.

With the examination proctoscope, a correct position of the operation area is set by pushing a depth setting piston, that is part of the handle, towards the skin when the proctoscope is aligned with the dentate line. The handle is then transferred to the MD, which is inserted into the rectum until the depth- setting piston touches the skin, ensuring a correct position of the operation area.

The MD have three operation areas that are positioned alongside the device at 3, 7, and 11 o'clock, which corresponds with the position of the three major internal hemorrhoids. Each operation area consists of 5 indentations, 4 smaller and one larger furthest in. The floor of the indentations has small holes, so when vacuum suction is applied within the device, the mucosa is sucked down into the indentations and thereby folding the mucosa above the hemorrhoids. A double needle is then pushed through the folded mucosa and docks with the ends of a loop of a suture that is stored in the suture cassette at the tip the tip of the device. When the needles are retracted, a loop of suture is introduced through the folded mucosa. The position of the sutures starts 10mm above the dentate line thanks to the settings done through the examination proctoscope and the depth setting piston. The sensation of pain is not present 10mm above the dentate line, which enables surgery without anesthesia. The stitches are 4mm wide, 3mm deep and 10mm long in the first four stitches and 6mm deep and 12mm long in the final stitch furthest in. The unit forming the walls of the indentations is divided into three longitudinal parts. When a supportive tray is removed the unit falls apart into three pieces and is removed, leaving the suture in the mucosa. Knots are then applied with a knot pusher, which pulls the folded mucosa together and the hemorrhoids are lifted inwards. The compressed mucosa is estimated to create multiple adhesion points/scar tissues that fixate the hemorrhoid in the new elevated position, ensuring a long-lasting result after the suture is absorbed (60-90 days). A special mucosa spatula is used to push out any protruding mucosa to make extraction of the device easier without damaging the tissue.

Number of subjects: 31-35 patients

The SCI-Pex study will evaluate the safety and performance of PexyEazy on patients with hemorrhoids grade II and III. For safety reasons will the first 6-10 patients undergo the procedure under general anesthesia and then the procedure will be done on awake patients (25) with 1 week, 3 months and 1 years follow up with questionnaires and a clinical examination after 3 months and 1 year to document result.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Hemorrhoidal disease grade II and III
* American Society of Anesthesiologists (ASA) classification I-III.

Exclusion Criteria:

* Previous surgical treatment for hemorrhoids by all methods except rubber band ligation or sclerosing injection therapy within the last 3 years.
* Previous surgical treatment with rubber band ligation or injection therapy within the last 2 months.
* More than three surgical treatments with rubber band ligation or sclerosing injection therapy within the last 3 years.
* Under medication with immunosuppressive drugs and/or anticoagulant drugs (not including 75mg acetylsalicylic acid) and not able to interrupt the anticoagulant drug medication or replace it with low molecular weight heparin for 5 days.
* Have ulcerative colitis, Crohn's disease or other intestinal inflammatory disease or presence of inflamed or thickened mucosa of the rectum.
* Presence of anal fissure, anal stenosis, stricture, fistulas or ulcers in the rectal area.
* The rectum has not been prepared prior to the investigation with rectal enema and is contaminated with feces that cannot easily be removed.
* Have schizophrenia, untreated depression or other mental illness or conditions that may affect judgment, sensation of pain or inability to complete the follow-up.
* Under medication of morphine or other strong painkillers, not including paracetamol.
* Fecal incontinence (not including soiling due to hemorrhoidal disease), or conditions with impaired sensation in the rectal area or impaired function of the anal sphincter.
* Previous rectal radiation.
* Rectal cancer or previous surgery due to rectal cancer.
* Pregnancy
* Hypercoagulability disorders or diseases that result in increased risk of bleeding.
* Impaired immune system or condition that increases the risk of infection.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2026-04-28 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Surgical result | Directly after the surgical procedure
  Clinical evaluation that a proper mucopexy has been achieved above all three locations (3, 7 and 11 o'clock) and any signs of bleeding or other damage to the mucosa, which is documented by the surgeon and by photography.
Validation of device | Directly after the surgical procedure.
  The handling and performance of the device is validated through a questionnaire that the surgeon fills out after the procedure.
Registered duration of surgery | Directly after the surgical procedure.
  Duration of surgery (minutes)
Presence of pain | Directly after the surgical procedure.
  The patient fill in a questionnaire with a scale between 1 and 10, where 1 is no pain and 10 is the worst possible pain.
Need of anesthesia, pain relief or local anesthesia | Directly after the surgical procedure.
  The need for per-operative anesthesia and/or sedation and/or pain relied (morphine) and/or local anesthesia will be registered.
Per-operative complications | Directly after the surgical procedure.
  Adverse events (both complication and device malfunction) during or directly after the procedure, which will be registered by a questionnaires filled in by patient and surgeon.

SECONDARY OUTCOMES:
Use of pain relief drugs after surgery | 1 week, 3 months and 1 year after surgery
  The use of pain relief drugs (name of drug, dosage, number/day)
Pain after surgery | 1 week, 3 months and 1 year after surgery
  The patient fill in a questionnaire with a scale between 1 and 10, where 1 is no pain and 10 is the worst possible pain.
Post operative complications | 1 week, 3 months and 1 year after surgery
  Registration of any post-operative complications (fecal incontinence, anal stenosis, bleeding, perianal hematoma, urinary retention or incontinence, presence of infection/abscess and assessment by Clavien-Dindo classification).
Clinical outcome | 3 months and 1 year after surgery
  Evaluation of the rectum and anal canal 3 months after the procedure to register presence of complications and recurrence of the hemorrhoidal disease. The result is documented by the surgeon and by a photography of the mucosa.
Change of symptoms | Before the procedure, 1 week, 3 months and 1 year after the procedure.
  Change of hemorrhoid symptoms through a questionnaire called Hemorrhoidal Disease Symptom Score and Hemorrhoidal Disease Symptom Score (HDSS and HSS). The score can vary between 4-28.The higher the value, the more severe/worse symptoms.
Change in quality of life | Before the procedure, 3 months and 1 year after the procedure.
  Change in quality of life through a questionnaire called 36-Item Short Form Health Survey (SF-36). The score can vary between 0-100.The higher the value, the better quality of life.
Duration of sick-leave/unable to perform normal activities. | 1 week, 3 months and 1 year after surgery
  The patient fills in a questionnaire about how long and to what degree the patient needed sick-leave or were not able to perform normal activities (in case the patient does not work).

OTHER OUTCOMES:
Cost | 3 month and 1 year
  Calculate the total cost of the procedure including the cost for treatment of any complications, use of pain relief drugs and sick leave during the 3 month follow up period.

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Kressner, Dr, Principal Investigator — Norrtälje Sjukhus
Locations (3):
- Sweden (3):
  - Frölunda Specialistsjukhus, Frölunda
  - Norrtälje Sjukhus, Norrtälje
  - Capio kirurgkliniken, Sophiahemmet, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
If data from the study is to be used for meta-analysis or review articles it will be shared upon request.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: From the start of the study to the end of the study.
Access Criteria: E-mail to office@developeration.se for requesting information.

REFERENCES:
- [Result] Aigner F, Gruber H, Conrad F, Eder J, Wedel T, Zelger B, Engelhardt V, Lametschwandtner A, Wienert V, Bohler U, Margreiter R, Fritsch H. Revised morphology and hemodynamics of the anorectal vascular plexus: impact on the course of hemorrhoidal disease. Int J Colorectal Dis. 2009 Jan;24(1):105-13. doi: 10.1007/s00384-008-0572-3. Epub 2008 Sep 3. PMID 18766355
- [Result] Aigner F, Kronberger I, Oberwalder M, Loizides A, Ulmer H, Gruber L, Pratschke J, Peer S, Gruber H. Doppler-guided haemorrhoidal artery ligation with suture mucopexy compared with suture mucopexy alone for the treatment of Grade III haemorrhoids: a prospective randomized controlled trial. Colorectal Dis. 2016 Jul;18(7):710-6. doi: 10.1111/codi.13280. PMID 26787597
- [Result] Gupta PJ, Kalaskar S, Taori S, Heda PS. Doppler-guided hemorrhoidal artery ligation does not offer any advantage over suture ligation of grade 3 symptomatic hemorrhoids. Tech Coloproctol. 2011 Dec;15(4):439-44. doi: 10.1007/s10151-011-0780-7. Epub 2011 Oct 28. PMID 22033542